CLINICAL TRIAL: NCT01920334
Title: Effects of Zolpidem CR in Sleep and Clinical Outcomes of Patients in Cardiac Intensive Care Unit
Brief Title: Effects of Zolpidem CR® in Sleep and Heart Recovery in Cardiac Intensive Care Unit Patients
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Associação Fundo de Incentivo à Pesquisa (Other)
Collaborators: Conselho Nacional de Desenvolvimento Científico e Tecnológico (Other Government)
Responsible Party: Principal Investigator, Patrick Rademaker Burke, Sleep Medicine PhD Student, Associação Fundo de Incentivo à Pesquisa
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1442/11, Ethics Committee; CardioHE, AFIP (Other: AFIP)
Record Dates: First submitted 2013-08-07; First posted 2013-08-12 (Estimated); Last update posted 2013-08-12 (Estimated); Status verified 2013-08

CONDITIONS: Acute Coronary Syndrome; Sleep Deprivation
Keywords: coronary disease; heart diseases; enzymes; sleep; troponin; zolpidem
MeSH Terms: conditions — Acute Coronary Syndrome; Sleep Deprivation; Coronary Disease; Heart Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Zolpidem CR 12.5mg (Experimental): Patients receive zolpidem CR 12.5mg at bedtime from the first night on the Cardiac Intensive Care Unit until their discharge from the hospital
  Interventions: Drug: Zolpidem CR 12.5mg
- Placebo (Placebo Comparator): Patients receive placebo at bedtime from the first night on the Cardiac Intensive Care Unit until their discharge from the hospital
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Zolpidem CR 12.5mg — Patients will be given zolpidem CR 12.5mg each night for, at least, 3 consecutive nights, including the first night on the Cardiac ICU, when the undergo a full-night polysomnography
  Other Names: Stillnox CR 12.5mg
  Arms: Zolpidem CR 12.5mg
Drug: Placebo — Patients will receive placebo pills at night, according to their usual sleep time, from the first night on the Cardiac ICU, until their hospital discharge
  Arms: Placebo

SUMMARY:
A double blind, randomized, placebo-controlled study will be conducted in cardiac ICU patients who had been diagnosed with acute coronary syndrome, using a sleep promoting drug (zolpidem controlled release).

The study hypothesis is that sleeping better can improve the heart recovery in patients with a diagnosis of acute coronary syndrome.

DETAILED DESCRIPTION:
The environment of an Intensive Care Unit (ICU) is notoriously inhospitable to patients who experience a period of sleep deprivation (SD). Recent research has shown that SD, even in the short-term, may be related to echo and electrocardiographic changes that may potentially be predictors of cardiac arrhythmias.

The objective is to evaluate the effects of early treatment with zolpidem controlled release (CR®) compared to a placebo on clinical and polysomnographic parameters for patients in a cardiac ICU who had recently been diagnosed with acute coronary syndrome.

A double blind, randomized, placebo-controlled study will be conducted in cardiac ICU patients who had been diagnosed with acute coronary syndrome. The patients in group A will receive placebo and patients in group B will receive zolpidem CR® 12.5 mg from the first night of hospitalization until their discharge. Patients will undergo overnight full polysomnography on the first night in the ICU and will complete a sleep diary with a visual analogue scale to evaluate sleep quality in the morning after the first 3 nights of hospitalization. The results of the routine ICU laboratory tests including the serum levels of cardiac enzymes [troponin T and creatine kinase MB (CK-MB)] will be collected preceding the first dose of the drug/placebo, and then daily thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Patients from 18 to 75 years of age
* Diagnosis of acute coronary syndrome
* Capable of swallowing pills
* Capable of filling in the questionaires

Exclusion Criteria:

* Class IV heart failure according to the New York heart association functional class,
* Patients in a coma
* Patients receiving mechanical ventilation
* Patients who regularly use benzodiazepines or other medications for inducing sleep

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2013-07; Primary Completion 2013-10 (Estimated); Study Completion 2014-01 (Estimated)

PRIMARY OUTCOMES:
Sleep efficiency | 1 day - the first night
  A full-night polysomnography is conducted in the first night on the ICU

SECONDARY OUTCOMES:
Troponin T | Within the first 3 days after an acute coronary syndrome diagnosis
  The serum troponin T is measured previously of the intervention and daily for 3 consecutive days
Creatine-kinase MB | Within the first 3 days after an acute coronary syndrome diagnosis
  The serum creatine-kinase MB is measured previously of the intervention and daily for 3 consecutive days

OTHER OUTCOMES:
Sleep quality analogue visual scale | 3 consecutive mornings
  After receiving the drug or placebo at night, the next morning the patients fill in the sleep quality visual analogue scale
The Pittsburgh Sleep Quality Index | 1 day, before the intervention
  Before the patient receives the drug/placebo, he fills in the Pittsburgh Sleep Quality Index
Epworth Sleepiness Scale | 1 day, before the intervention
  Before receiving the drug or placebo at night, patients fill in the Epworth Sleepiness Scale
Insomnia Severity Index | 1 day, before the intervention
  Before receiving the drug or placebo at night, patients fill in the Insomnia Severity Index

CONTACTS AND LOCATIONS:
Overall Officials: Patrick R Burke, MD, Principal Investigator — Associação Fundo de Incentivo à Pesquisa
Locations (1):
- Hospital São Paulo, São Paulo, São Paulo, Brazil